CLINICAL TRIAL: NCT05899127
Title: Effects of Intravenous Lidocaine Infusion on Stress Response in Patients Undergoing Abdominal Surgery During Perioperative Anesthesia and Its Correlation With Serum Orphanin FQ (N/OFQ)
Brief Title: Relationship Between Lidocaine and Serum Orphanin FQ (N/OFQ)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Hospital of Shanxi Medical University (Other)
Responsible Party: Principal Investigator, Zheng Guo, Professor, Second Hospital of Shanxi Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: hanyi20230118
Record Dates: First submitted 2023-02-17; First posted 2023-06-12 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Stress Reaction
MeSH Terms: conditions — Fractures, Stress | interventions — Lidocaine; Sufentanil; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lidocaine (Experimental): Lidocaine will be injected intravenously at 1.5mg/kg during anesthesia induction and intravenously pumped at 1.5mg/kg/h during anesthesia induction.
  Interventions: Drug: Lidocaine
- Control group (Placebo Comparator): Normal saline will be injected intravenously at 1.5mg/kg during the induction period and intravenously pumped at 1.5mg/kg/h during the induction period.
  Interventions: Drug: 0.9%NaCl

INTERVENTIONS:
Drug: Lidocaine — 1.5mg/kg induction，1.5 mg/kg/h maintenance
  Other Names: Sufentanil,Etomidate,Rocuronium,Propofol,Remifentanil
  Arms: Lidocaine
Drug: 0.9%NaCl — 2mg/kg induction，1.5 mg/kg/h maintenance
  Other Names: Sufentanil,Etomidate,Rocuronium,Propofol,Remifentanil
  Arms: Control group

SUMMARY:
The intravenous injection of lidocaine during the perioperative period has been widely used in various types of surgeries. Its clinical effect includes reducing stress response during anesthesia, decreasing pain and opioid consumption, lowering the incidence of postoperative nausea, vomiting, cognitive dysfunction, and reducing the injection pain of propofol. However, despite the positive impact of lidocaine on surgical patients, its mechanism of action remains unclear. Serum N/OFQ is a neurotransmitter that plays an important role in regulating pain and emotion. Therefore, this study aims to explore the effects of perioperative intravenous injection of lidocaine on stress responses in surgical patients, as well as its mechanism of action, and whether Serum N/OFQ participates in this process.

DETAILED DESCRIPTION:
We hypothesize that intravenous injection of lidocaine during the perioperative period can reduce expression of endogenous opioid peptides, which in turn can decrease secretion of IL-6 and TNF-α, ultimately leading to a reduction in perioperative stress response. This randomized controlled trial will be conducted at the Second Hospital of Shanxi Medical University in China, with the aim of observing changes in stress-related indicators (blood pressure, heart rate, heart rate variability, IL-6, TNF-α, as well as Serum N/OFQ ) between patients undergoing abdominal surgery under total intravenous general anesthesia with and without lidocaine injection. Lidocaine will be administered as a loading dose during anesthesia induction and continued via infusion until the end of anesthesia maintenance, with appropriate depth of anesthesia or BIS readings utilized for monitoring anesthesia depth. Routine monitoring parameters, including blood pressure, heart rate, SpO2, and electrocardiogram, will be recorded and analyzed. Blood samples will be collected 30 minutes before anesthesia induction, 1 minute after tracheal intubation, and at the end of surgery. The use of lidocaine will be evaluated for its impact on perioperative stress response in patients undergoing abdominal surgery, with the relationship to changes in levels of endogenous opioid peptides explored.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II
* Patients undergoing elective abdominal surgery with anesthesia duration less than 1-2h

Exclusion Criteria:

* It is estimated that patients with difficulty in tracheal intubation (poor head and neck mobility, history of airway surgery, history of OSAHS, nail to chin distance<6cm, Malampati grade 3 and above, mouth opening<2.5cm, obesity (BMI>30kg · m-2), etc.)
* Hypertension patients (clinically diagnosed as hypertension), coronary heart disease patients (with typical symptoms of angina pectoris and exclusion of aortic valve disease, clear history of old myocardial infarction, clear history of acute myocardial infarction)
* Patients with diabetes and central nervous system diseases
* Patients with long-term use of sedatives or antidepressants
* Patients with a history of alcoholism or drug dependence
* Asthma or reactive airway disease
* Shock, severe hypotension, severe arrhythmia and other adverse events occurred during the operation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-07-22 (Actual); Primary Completion 2024-07-30 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Stress response index | 24 hours
  It includes blood pressure, heart rate, heart rate variability,IL-6 and TNF-α.
Serum Norepinephrine | 24 hours
  It may have been involved in the regulation of stress response processes by lidocaine.

CONTACTS AND LOCATIONS:
Locations (1):
- Second of Shanxi Medical University, Taiyuan, Shanxi, China